CLINICAL TRIAL: NCT02877225
Title: A Single-Dose, Open-Label, Randomized, Replicate Crossover Study in Healthy Adult Subjects to Assess the Bioequivalence of an Ibrutinib 140-mg Tablet Compared to the IMBRUVICA 140-mg Capsule
Brief Title: Study to Assess the Bioequivalence of Ibrutinib 140 Milligram (mg) Tablet to 140 mg IMBRUVICA Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR108174; 54179060CLL1022 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Healthy
MeSH Terms: interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence 1 : ABAB (Experimental): Participants will receive 140 milligram (mg) of ibrutinib administered as one IMBRUVICA 140-mg oral capsule (Treatment A) in Period 1, 140 mg of ibrutinib administered as one ibrutinib 140-mg oral tablet (Treatment B) in Period 2, then Treatment A in period 3 and then followed by Treatment B in Period 4. Each intervention Period will be separated by a washout period of 7-9 days.
  Interventions: Drug: Ibrutinib; Drug: IMBRUVICA
- Treatment Sequence 2 : BABA (Experimental): Participants will receive (Treatment B) Period 1, then Treatment A in Period 2, then Treatment B in Period 3 and then followed by Treatment A in Period 4. Each intervention Period will be separated by a washout period of 7-9 days.
  Interventions: Drug: Ibrutinib; Drug: IMBRUVICA

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib (test treatment) 140 milligram (mg), tablet.
Drug: IMBRUVICA — IMBRUVICA (reference treatment), 140-mg capsule
  Other Names: Ibrutinib

SUMMARY:
The purpose of this study is to demonstrate the bioequivalence (BE) of a new formulation of ibrutinib to the marketed Imbruvica formulation in healthy adults under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Be a man or woman between 18 and 55 years of age, inclusive, at screening
* If a woman, must have a negative serum beta human chorionic gonadotropin (Beta - hCG) pregnancy test at screening and on Day -1 of each treatment period
* Body Mass Index (BMI); weight [kilogram (kg)]/height^2 [meter(m)^2)] between 18.0 and 30.0 kg/m2 (inclusive) and body weight not less than 50 kg at screening
* If a woman, must be of nonchildbearing potential, defined as either: a) Postmenopausal : A postmenopausal state is defined as no menses for at least 12 months without an alternative medical cause and a serum follicle stimulating hormone (FSH) level in the postmenopausal range (greater (>)40 International Units Per Liter (IU/L) or milli-international units per milliliter(mIU/mL), OR, b) Permanently sterile: Permanent sterilization methods include subtotal or total hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures (without reversal operation), bilateral oophorectomy, and transcervical sterilization
* Blood pressure (supine after at least 5 minutes rest) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic at screening
* Alanine aminotransferase, aspartate aminotransferase (AST), alkaline phosphatase (ALP) and total bilirubin equal to or lower than the upper limit of normal (per National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [CTCAE]) at screening

Exclusion Criteria:

* History of current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the Investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology or biochemistry at screening as deemed appropriate by the Investigator
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG) at screening as deemed appropriate by the Investigator
* History of clinically significant allergies, especially known hypersensitivity or intolerance to sulfonamide or beta-lactam antibiotics
* Positive test for hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies at screening
* Positive test for human immunodeficiency virus type 1 (HIV-1) or HIV-2 antibodies at screening
* Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 1 month or within a period less than 10 times the drug's half-life, whichever is longer, before the planned first intake of study drug
* History of clinically significant allergies, especially known hypersensitivity or intolerance to sulfonamide or beta-lactam antibiotics

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2016-11-11 (Actual)

PRIMARY OUTCOMES:
Area Under Concentration from time zero to the last quantifiable (AUC [0-last]) | Predose up to Day 3
  Area under the concentration-time curve (AUC) from time 0 to the time of the last measurable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Predose up to Day 3
  The AUC (0-infinity) is the area under the plasma concentration time curve from time zero to infinite time, calculated as the sum of AUC (0-last) and C (0-last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant.
Maximum Observed Analyte Concentration (Cmax) | Predose up to Day 3
  Maximum observed analyte concentration will be assessed.
Time to Reach Maximum Concentration (Tmax) | Predose up to Day 3
  Tmax is defined as actual sampling time to reach maximum observed analyte concentration will be assessed.
Apparent Terminal Elimination Halflife (t1/2term) | Predose up to Day 3
  The elimination halflife (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration time curve and calculated as 0.693/apparent terminal elimination rate constant (λz).
Apparent Terminal Elimination Rate Constant (lambda z) | Predose up to Day 3
  Apparent terminal elimination rate constant, estimated by linear regression using the terminal loglinear phase of the log transformed concentration versus time data.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Approximately 59 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tempe, Arizona, United States